CLINICAL TRIAL: NCT00526955
Title: Duration and Force Variations in Applied Kinesiology Manual Muscle Testing
Status: Completed | Type: Observational
Sponsor: Logan College of Chiropractic (Other)
Other Study IDs: RD0827070108
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: Manual muscle testing

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To investigate the effect of duration of Applied Kinesiology manual muscle testing on "strong" versus "weak" result of the test.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* willing to participate

Exclusion Criteria:

* Major injury or conditions which would prevent muscle testing of the shoulder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-11; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Force over time during a manual muscle test and a maximal voluntary isometric contraction | 1 to 6 seconds

SECONDARY OUTCOMES:
Facilitated (strong) or inhibited (weak) rating of muscle | 1 to 6 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Katharine M Conable, D.C., Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States